CLINICAL TRIAL: NCT04489706
Title: A Clinical Trial to Evaluate the Efficacy, Safety, and Tolerability of Arsenic Trioxide for Injection in Patients With Recurrent and Metastatic Ovarian Cancer and Endometrial Cancer With P53 Mutation
Brief Title: Arsenic Trioxide in Recurrent and Metastatic Ovarian Cancer and Endometrial Cancer With P53 Mutation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2020)96
Record Dates: First submitted 2020-07-05; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: Arsenic Trioxide for injection; P53 mutation; Recurrent and Metastatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Arsenic Trioxide; Injections; Long-Term Synaptic Depression

STUDY DESIGN:
Intervention Model Description: Histologically confirmed ovarian cancer and endometrial cancer patients with P53 mutation who had relapsed or metastasized after at least one line of standard system therapy. 20 subjects will be enrolled in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- P53 mutation arm (Experimental): patients of recurrent and metastatic ovarian cancer and endometrial cancer associated with P53 mutation
  Interventions: Drug: Arsenic trioxide for injection

INTERVENTIONS:
Drug: Arsenic trioxide for injection — Arsenic trioxide for injection, 0.16 mg/kg (maximum single dose is 10 mg), daily IV drip, d1 to d14, once every 28 days, for six cycles of treatment or until one of the following events occurs: Initiation of new anti-tumor therapy, disease progression, withdrawal of Informed consent form (ICF) and/or death.
  Other Names: Arsenic trioxide for injection，producted by Beijing SL Pharmaceutical Co., Ltd.

SUMMARY:
This study is a Single-center, open, single-arm and non-randomized clinical trial in China. The aim of this study is to evaluate the efficacy, safety, and tolerability of Arsenic trioxide for injection in patients with recurrent and metastatic ovarian cancer and endometrial cancer with P53 mutation A group of 20 women with histologically confirmed ovarian cancer and endometrial cancer who had previously received at least one line of standard system therapy and had relapsed or metastasized had a P53 mutation.

The subjects of this study are histologically confirmed ovarian cancer and endometrial cancer patients with P53 mutation who had relapsed or metastasized after at least one line of standard system therapy. 20 subjects will be enrolled in this study.

Main objectives of the study are Independent imaging and tumor markers assess ORR (objective response rate) in patients with recurrent and metastatic ovarian cancer and endometrial cancer with P53 mutation treated with Arsenic trioxide for injection, based on RECIST v1.1 （Response evaluation criteria in solid tumors） Secondary objectives including DCR (Disease control rate), CBR (Clinical benefit rate), PFS (Progression free survival), OS (Overall survival), DoR (Duration of response), safety and tolerability of Arsenic trioxide for injection, based on NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events), evaluated by researchers and life quality.

The study will be conducted in the department of obstetrics and gynecology in Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital.

Research intervention: injection Arsenic trioxide, 0.16mg/kg (maximum single dose is 10 mg), daily IV drip, d1 to d14, once every 28 days, for six cycles of treatment or until one of the following events occurs: Initiation of new anti-tumor therapy, disease progression, withdrawal of Informed consent form (ICF) and/or death.

The duration of this study will be 2.5 years; the admission period will be 1.5 years and the follow-up period will be 1 year.

DETAILED DESCRIPTION:
The P53 mutation plays an important role in the development of ovarian cancer and endometrial cancer, which has been found to occur in more than 95% of high grade serous ovarian cancers, 25% of the endometrial cancer, with serous endometrial cancer having a P53 mutation rate of 88%.

In Acute promyelocytic leukemia treatment, a combination of retinoic acid (ATRA) and Arsenic trioxide (ATO) has an extremely high cure rate, with an overall five-year survival rate of 88% , the therapeutic effect of ATO on some hematologic malignancies has been widely recognized. What's more, it is also found that arsenic has potential therapeutic effects on a variety of solid tumors, including Esophageal, liver and lymphoma.

Preciously research modified H1299 cells with structural mutant P53 (p53-R175H) and treated them with doxcycline to knock down p53-R175H. The system was able to determine whether the observed antitumor effects were dependent on the structural mutant p53. In the transplanted tumor model of this cell line in mice, ATO significantly inhibited the tumor growth rate. In mice fed with doxcycline, cancer cells expressed almost no P53-R175H, and the ATO had limited inhibitory effect on the transplanted tumor model. These results suggest that ATO inhibits tumor cell proliferation mainly by targeting structural mutant p53.

Researchers tested the antineoplastic effects of ATO on various solid tumor PDX models on a small scale. the results showed than the antineoplastic effect of ATO on the PDX (Patient-Derived tumor Xenograft) model was observed in several solid tumor models with structural mutant P53, including liver, Lung, and Pancreatic Cancer. This suggests that the antineoplastic effects of ATO are not limited to the types of cancer. Its anti-tumor effect is only related to the structural mutant p53 in cancer cells.

Previous studies have shown that Arsenic trioxide can bind to the structural mutant P53 and partially restore its function, so the goal of this study is to observe the efficacy, safety, and tolerability of Arsenic trioxide for injection in patients with recurrent and metastatic ovarian cancer and endometrial cancer combined with P53 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants (or their legal Representatives/guardians) are required to sign an informed consent form, indicating that they understand the objectives of the study, necessary procedures and are willing to participate in the study.
* Women over 18 years of age with histologically confirmed recurrence or metastasis of ovarian cancer or endometrial cancer.
* Laboratory confirmed P53 Gene Mutation.
* Previously received no less than 1-line treatment in the past with disease recurrence or progression.
* Disease Recurrence or progression (based on clinical, tumor markers, or imaging findings) occurs less than 6 months after the last treatment.
* At least one measurable lesion was confirmed by independent central imaging, according to RECIST V1.1, or elevation of tumor markers.
* ECOG PS (Eastern Cooperative Oncology Group Performance Status) score 0-1
* Estimated survival time ≥12 weeks.
* Sexually active, fertile subjects and their spouses have to agree to contraception throughout the study and within 90 days of the last study drug being given.

Exclusion Criteria:

* Hematopoiesis or organ dysfunction (blood products, such as blood transfusions, should not be used until less than 14 days before the first dose of the drug is studied) .
* ANC (Absolute neutrophil count）<1.5×10^9/L.
* HGB（Hemoglobin）< 8 g/dL.
* PLT (Platelet）<100×10^9/L.
* TBIL (Total bilirubin）>1.5 × ULN（Upper limit of normal)
* AST（Aspartate transferase）and/or ALT（Alanine aminotransferase）>3 × ULN，>5 × ULN in subjects with liver metastases.
* Cr (Creatine) >1.5 × ULN.
* INR (International normalized ratio)>1.5 × ULN，aPTT (activated Partial thromboplastin time) >1.5 × ULN, (INR is only applicable to subjects who have not received anticoagulation therapy).
* Radiation therapy less than 4 weeks before the first dose of study drug, or chemotherapy, biotherapy, endocrine therapy or small molecule targeted therapy before the first dose of study drug (elution ≥5 half-lives can be grouped).
* Toxic response to previous antitumor therapy has not yet recovered to 1 grade, according to NCI CTCAE V5.0, except for alopecia.
* Clinically significant active infection.
* Clinically significant active bleeding.
* Alcoholism or drug addiction.
* A history of clinically significant liver disease, including active viral or other hepatitis, alcohol abuse, or cirrhosis, except in subjects with a prior hepatitis which is inactive, confirmed by PCR (Polymerase chain reaction).
* HIV (Human immunodeficiency virus) infection.
* NYHA (The New York Heart Association) Class II or above Heart failure; History of myocardial infarction or unstable Angina within 6 months before treatment; History of myocardial infarction or unstable angina within 6 months before treatment.
* Pregnancy, breastfeeding or planning to become pregnant during the study period.
* Bowel obstruction within 12 weeks before the first dose of the drug.
* Received major surgery within 4 weeks before the first dose of the study drug.
* Received oral or intravenous Glutathione within 3 weeks before the start of treatment.
* Known to be allergic or hypersensitive to any ingredient of Arsenic trioxide.
* Subjects with poor adherence, or with any unsuitability to participate in this trial; Subjects with any clinical or laboratory abnormalities were not eligible to participate in this clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients woth ovarian cancer or endometrial cancer.
Enrollment: 20 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
the diameter of the measurable lesion | From the date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, through study completion, an average of 1 year.
  The retraction degree of the lesion which was detected in the beginning of the study (measured by CT, MRI or ultrasound).
the level of tumor markers in serum. | From the date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, through study completion, an average of 1 year.
  the level of CA125 (carbohydrate antigen 125), HE4 (human epididymis protein 4) or other abnormal tumor markers in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Feng, PhD, Study Chair — Ruijin Hospital
Locations (1):
- Shanghai JiaoTong University School of Medicine affliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zehir A, Benayed R, Shah RH, Syed A, Middha S, Kim HR, Srinivasan P, Gao J, Chakravarty D, Devlin SM, Hellmann MD, Barron DA, Schram AM, Hameed M, Dogan S, Ross DS, Hechtman JF, DeLair DF, Yao J, Mandelker DL, Cheng DT, Chandramohan R, Mohanty AS, Ptashkin RN, Jayakumaran G, Prasad M, Syed MH, Rema AB, Liu ZY, Nafa K, Borsu L, Sadowska J, Casanova J, Bacares R, Kiecka IJ, Razumova A, Son JB, Stewart L, Baldi T, Mullaney KA, Al-Ahmadie H, Vakiani E, Abeshouse AA, Penson AV, Jonsson P, Camacho N, Chang MT, Won HH, Gross BE, Kundra R, Heins ZJ, Chen HW, Phillips S, Zhang H, Wang J, Ochoa A, Wills J, Eubank M, Thomas SB, Gardos SM, Reales DN, Galle J, Durany R, Cambria R, Abida W, Cercek A, Feldman DR, Gounder MM, Hakimi AA, Harding JJ, Iyer G, Janjigian YY, Jordan EJ, Kelly CM, Lowery MA, Morris LGT, Omuro AM, Raj N, Razavi P, Shoushtari AN, Shukla N, Soumerai TE, Varghese AM, Yaeger R, Coleman J, Bochner B, Riely GJ, Saltz LB, Scher HI, Sabbatini PJ, Robson ME, Klimstra DS, Taylor BS, Baselga J, Schultz N, Hyman DM, Arcila ME, Solit DB, Ladanyi M, Berger MF. Mutational landscape of metastatic cancer revealed from prospective clinical sequencing of 10,000 patients. Nat Med. 2017 Jun;23(6):703-713. doi: 10.1038/nm.4333. Epub 2017 May 8. PMID 28481359
- [Result] Yang WL, Gentry-Maharaj A, Simmons A, Ryan A, Fourkala EO, Lu Z, Baggerly KA, Zhao Y, Lu KH, Bowtell D, Jacobs I, Skates SJ, He WW, Menon U, Bast RC Jr; AOCS Study Group. Elevation of TP53 Autoantibody Before CA125 in Preclinical Invasive Epithelial Ovarian Cancer. Clin Cancer Res. 2017 Oct 1;23(19):5912-5922. doi: 10.1158/1078-0432.CCR-17-0284. Epub 2017 Jun 21. PMID 28637689
- [Result] Schultheis AM, Martelotto LG, De Filippo MR, Piscuglio S, Ng CK, Hussein YR, Reis-Filho JS, Soslow RA, Weigelt B. TP53 Mutational Spectrum in Endometrioid and Serous Endometrial Cancers. Int J Gynecol Pathol. 2016 Jul;35(4):289-300. doi: 10.1097/PGP.0000000000000243. PMID 26556035
- [Result] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Result] Soragni A, Janzen DM, Johnson LM, Lindgren AG, Thai-Quynh Nguyen A, Tiourin E, Soriaga AB, Lu J, Jiang L, Faull KF, Pellegrini M, Memarzadeh S, Eisenberg DS. A Designed Inhibitor of p53 Aggregation Rescues p53 Tumor Suppression in Ovarian Carcinomas. Cancer Cell. 2016 Jan 11;29(1):90-103. doi: 10.1016/j.ccell.2015.12.002. Epub 2015 Dec 31. PMID 26748848
- [Result] Leijen S, van Geel RM, Sonke GS, de Jong D, Rosenberg EH, Marchetti S, Pluim D, van Werkhoven E, Rose S, Lee MA, Freshwater T, Beijnen JH, Schellens JH. Phase II Study of WEE1 Inhibitor AZD1775 Plus Carboplatin in Patients With TP53-Mutated Ovarian Cancer Refractory or Resistant to First-Line Therapy Within 3 Months. J Clin Oncol. 2016 Dec 20;34(36):4354-4361. doi: 10.1200/JCO.2016.67.5942. Epub 2016 Oct 28. PMID 27998224
- [Result] Martins CP, Brown-Swigart L, Evan GI. Modeling the therapeutic efficacy of p53 restoration in tumors. Cell. 2006 Dec 29;127(7):1323-34. doi: 10.1016/j.cell.2006.12.007. Epub 2006 Dec 21. PMID 17182091
- [Result] Ventura A, Kirsch DG, McLaughlin ME, Tuveson DA, Grimm J, Lintault L, Newman J, Reczek EE, Weissleder R, Jacks T. Restoration of p53 function leads to tumour regression in vivo. Nature. 2007 Feb 8;445(7128):661-5. doi: 10.1038/nature05541. Epub 2007 Jan 24. PMID 17251932
- [Result] Xue W, Zender L, Miething C, Dickins RA, Hernando E, Krizhanovsky V, Cordon-Cardo C, Lowe SW. Senescence and tumour clearance is triggered by p53 restoration in murine liver carcinomas. Nature. 2007 Feb 8;445(7128):656-60. doi: 10.1038/nature05529. Epub 2007 Jan 24. PMID 17251933
- [Result] Abaza Y, Kantarjian H, Garcia-Manero G, Estey E, Borthakur G, Jabbour E, Faderl S, O'Brien S, Wierda W, Pierce S, Brandt M, McCue D, Luthra R, Patel K, Kornblau S, Kadia T, Daver N, DiNardo C, Jain N, Verstovsek S, Ferrajoli A, Andreeff M, Konopleva M, Estrov Z, Foudray M, McCue D, Cortes J, Ravandi F. Long-term outcome of acute promyelocytic leukemia treated with all-trans-retinoic acid, arsenic trioxide, and gemtuzumab. Blood. 2017 Mar 9;129(10):1275-1283. doi: 10.1182/blood-2016-09-736686. Epub 2016 Dec 21. PMID 28003274
- [Result] Zhang TD, Chen GQ, Wang ZG, Wang ZY, Chen SJ, Chen Z. Arsenic trioxide, a therapeutic agent for APL. Oncogene. 2001 Oct 29;20(49):7146-53. doi: 10.1038/sj.onc.1204762. PMID 11704843
- [Derived] Tang Y, Song H, Wang Z, Xiao S, Xiang X, Zhan H, Wu L, Wu J, Xing Y, Tan Y, Liang Y, Yan N, Li Y, Li J, Wu J, Zheng D, Jia Y, Chen Z, Li Y, Zhang Q, Zhang J, Zeng H, Tao W, Liu F, Wu Y, Lu M. Repurposing antiparasitic antimonials to noncovalently rescue temperature-sensitive p53 mutations. Cell Rep. 2022 Apr 12;39(2):110622. doi: 10.1016/j.celrep.2022.110622. PMID 35417717